CLINICAL TRIAL: NCT01439178
Title: Acute Changes in Intraocular Cytokines After Intravitreal Bevacizumab
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Won Ki Lee, Preofessor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC11MISI0391
Record Dates: First submitted 2011-08-29; First posted 2011-09-23 (Estimated); Last update posted 2011-09-23 (Estimated); Status verified 2011-09

CONDITIONS: Complications of Diabetes Mellitus
MeSH Terms: conditions — Diabetes Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intravitreal Avastin Day 2 (Experimental): randomized to either treatment with preoperative IVB 2 days before PPV (Group A) or 7 days before PPV (Group B).
  Interventions: Drug: Intravitreal Avastin injection
- Intravitreal Avastin Day 7 (Active Comparator): randomized to either treatment with preoperative IVB 2 days before PPV (Group A) or 7 days before PPV (Group B).
  Interventions: Drug: Intravitreal Avastin injection

INTERVENTIONS:
Drug: Intravitreal Avastin injection — Bevacizumab (1.25 mg in 0.05 ml) (Avastin; Genentech Inc., San Francisco, CA, USA) will be injected through the pars plana at 3.5 mm from the limbus, using 30 gauge needle.

SUMMARY:
Purpose: To evaluate the acute changes in intraocular cytokines after intravitreal bevacizumab (IVB) in proliferative diabetic retinopathy.

Design: Prospective, open-label, controlled, randomized interventional clinical trial.

Participants: Twenty eyes of 28 consecutive patients who are scheduled for pars plana vitrectomy (ppV) for proliferative diabetic retinopathy were prospectively enrolled.

Methods: All patients were randomly assigned to receive IVB either at 2 or 7 days before ppV. Aqueous humor samples were taken from anterior chamber just before IVB and at the time of surgery. Multiplex cytokine array were used to assay various cytokines

ELIGIBILITY:
Inclusion Criteria:

* Patients with proliferative diabetic retinopathy who were scheduled for PPV for vitreous hemorrhage or tractional retinal detachment (TRD)

Exclusion Criteria:

* Eyes with any pharmacologic intervention on study eye within 6 months
* Eyes with panretinal photocoagulation on study eye within 3 months
* Eyes with any pharmacologic intervention on fellow eye within 3 months,
* History of ocular diseases other than diabetic retinopathy
* History of PPV on study eye
* History of systemic thromboembolic events including myocardial infarction and cerebrovascular accidents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-11 (Estimated); Study Completion 2011-11 (Estimated)

PRIMARY OUTCOMES:
intraocular VEGF levels (pg/ml) in both groups (measured in aqueous humor), using multiplex beads immunoassay | At day 2 after IVB in Group 1, day 7 after IVB at group 2.
  Because we want to compare the differences between day 2 and day 7, vitrectomy will be performed at day 2 in group 1 and day 7 in group 2.
  That's why the time frame has two time point

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul Saint Mary's hospital, Seoul, Seoul, South Korea